CLINICAL TRIAL: NCT00695006
Title: Manual Therapy, Exercise and Traction for Patients With Cervical Radiculopathy: A RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rocky Mountain University of Health Professions (Other)
Responsible Party: Ian Young, Advance Rehab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5388642
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2008-06-25 (Estimated); Status verified 2008-06

CONDITIONS: Cervical Radiculopathy
Keywords: manual therapy, cervical traction, cervical radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — Traction

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- II (Sham Comparator): Sham Traction
  Interventions: Other: Sham Traction
- I (Active Comparator): Traction
  Interventions: Other: Traction

INTERVENTIONS:
Other: Sham Traction — Traction <5lbs
  Arms: II
Other: Traction — Standard supine intermittent traction
  Arms: I

SUMMARY:
To date, optimal strategies for the management of patients with Cervical Radiculopathy (CR) remain elusive. The purpose of this study was to compare the effects of manual therapy, exercise, and cervical traction to manual therapy, exercise, and sham traction on pain, function and disability in patients with CR.

ELIGIBILITY:
Inclusion Criteria:

* 3 of 4 positive on CPR, 18-70yrs

Exclusion Criteria:

* history of previous cervical or thoracic spine surgery
* bilateral upper extremity symptoms
* signs or symptoms of UMN disease
* medical "red flags"(tumor, fracture, rheumatoid arthritis, osteoporosis, prolonged steroid use)
* cervical spine injections (steroidal) in the past two weeks
* current use of steroidal medication prescribed for their radiculopathy symptoms

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index | 2wk, 4wk, 3mo, 6mo
Patient Specific Functional Scale | 2wk, 4wk, 3mo, 6mo
Numeric Pain Rating Scale | 2wk, 4wk, 3mo, 6mo

SECONDARY OUTCOMES:
Global Rating Of Change | 2wk, 4wk, 3mo, 6mo
Body Diagram | 2wk, 4wk, 3mo, 6mo
Fear Avoidance Belief Questionnaire | 2wk, 4wk, 3mo, 6mo
Satisfaction | 2wk, 4wk, 3mo, 6mo
Grip Strength | 2wk, 4wk

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Young, PT, Principal Investigator — Advance Rehab at Fredericksburg Orthopaedics
Locations (1):
- Advance Rehab at Fredericksburg Orthopaedics, Fredericksburg, Virginia, United States